CLINICAL TRIAL: NCT03070808
Title: The Influence of Significant Weight Lost on the Quality of Voice
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Dr Oded Cohen, Doctor, Kaplan Medical Center
Other Study IDs: 0005-17-KMC
Record Dates: First submitted 2017-02-21; First posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-02

CONDITIONS: Obesity, Morbid; Voice Alteration
Keywords: obesity; voice
MeSH Terms: conditions — Obesity, Morbid; Dysphonia; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rate of obesity and bariatric surgery is rising steadily. Though Bariatric Surgery Influences on aspects such as endocrin analysis, finance, etc are well tested, quantitative and quality voice impacts have not been evaluated. The aim of the study is to recruit 50 patients who underwent bariatric surgery and compare voice quality in each of these patients before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese
* Candidates for bariatric Surgery

Exclusion Criteria:

* History of benign \ malignant disease of the larynx.
* History of head and neck tumors
* History of radiation therapy of the neck
* BMI under 30 pre-surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, 18 years and over, entended for Bariatric Surgery at Kaplan Medicle Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-03-15 (Estimated); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
Stroboscopic evaluation of the larynx | 2/16-2/20
  A visual examination of the larynx

SECONDARY OUTCOMES:
Dysphagia handicap Index | 2/16-2/20
  Validitated questioners for dysphagia which result in a score
EAT 10 | 2/16-2/20
  Validitated questioners for dysphagia which result in a score
Voice Handicap Index | 2/16-2/20
  Validitated questioners for dysphagia which result in a score
Average Fundamental frequency | 2/16-2/20
  part of voice assessment, in Hertz
Mean Fundamental frequency | 2/16-2/20
  part of voice assessment, in Hertz
Highest Fundamental frequency | 2/16-2/20
  part of voice assessment, in Hertz
Lowest Fundamental frequency | 2/16-2/20
  part of voice assessment, in Hertz
Standard deviation of Fundamental frequency | 2/16-2/20
  part of voice assessment, in numbers
Noise to harmonic ratio | 2/16-2/20
  part of voice assessment, a descripitive measure of voice quality
Voice turbulence Index | 2/16-2/20
  part of voice assessment
Absolute gitter | 2/16-2/20
  Variability of frequency
Jitter percent | 2/16-2/20
  assessment of voice variability
Shimmer percent | 2/16-2/20
  assessment of voice variability
Shimmer in dB | 2/16-2/20
  variability of voice volume

IPD SHARING:
Plan to Share IPD: Undecided